CLINICAL TRIAL: NCT05539118
Title: Interferon-α1b (IFN-α1b) Combined With Toripalimab and Anlotinib Hydrochloride in Patients With Advanced Unresectable Melanoma
Brief Title: Interferon-α1b Combined With Toripalimab and Anlotinib Hydrochloride in Advanced Unresectable Melanoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20222092-C-1
Record Dates: First submitted 2022-08-17; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Melanoma
Keywords: Melanoma; unresectable; Interferon-alfa1b; Toripalimab; Anlotinib
MeSH Terms: conditions — Melanoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human interferon α1b + toripalimab + anlotinib hydrochloride (Experimental): Recombinant human interferon α1b administered 600μg every other day. Toripalimab administered 240mg intravenously every three weeks. Anlotinib hydrochloride given 12mg or 10mg or 8mg orally (Daily for two weeks continuously, followed by one week of rest). A recommended phase II dose (RP2D) of anlotinib hydrochloride will be determined.
  Interventions: Drug: Recombinant human interferon α1b; Drug: Toripalimab; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Recombinant human interferon α1b — Recombinant human interferon α1b is a protein with potent antiviral, antiproliferative and immunomodulatory properties.
Drug: Toripalimab — Toripalimab is a recombinant, humanized programmed death receptor (PD-1) monoclonal antibody that binds to PD- and prevents binding of PD-1 with programed death ligands 1 (PD-L1) and PD-L2. It can function to activate cytotoxic T lymphocytes and inhibit tumor growth.
Drug: Anlotinib hydrochloride — Anlotinib hydrochloride is a novel oral tyrosine kinase inhibitor (TKI) targeting vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR) and c-kit.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant human interferon-α1b (IFN-α1b) combined with toripalimab and anlotinib hydrochloride in patients with unresectable advanced melanoma. This study consists of 2 phases（ Ib / II）. Phase Ib will determine the recommended phase Ⅱ dose for anlotinib hydrochloride. Phase II will evaluate the efficacy and safety of the triple combination regimens.

DETAILED DESCRIPTION:
This is a single-arm, single-center Phase Ib/II trial to evaluate the efficacy and safety of the combination of recombinant human interferon α1b plus toripalimab and anlotinib hydrochloride in patients with unresectable Stage IIIc, Stage IIId, and Stage IV melanoma(AJCC 8th). Phase I is to evaluate the dose-limiting toxicities (DLT) and determine the recommended Phase II dose (RP2D) of anlotinib hydrochloride in patients with unresectable advanced melanoma receiving recombinant human interferon α1b 600ug QOD plus toripalimab 240mg Q3W. Anlotinib hydrochloride will be given in a dose descending manner(12mg- 10mg- 8mg). In the phase II study, 30 Phase II will enroll 30 patients. The primary endpoint in the II phase is objective response rate (ORR) and progression-free survival (PFS). The second endpoint is disease control rate (DCR), clinical benefit rate (CBR), duration of response (DOR), and overall survival(OS). The safety profile of this combined IFN-α1b/ toripalimab/anlotinib hydrochloride regimen will be monitored during both phases. Specifically, phase Ib will evaluate dose-limiting toxicities(DLT). Phase II will evaluate the numbers and severity of toxicity per the Criteria for Adverse Events version 5 (CTCAEv) including but not limited to all adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75.
2. ECOG performance status of 0 or 1
3. Life expectancy ≥ 3 months;
4. Histologically or cytologically confirmed diagnosis of unresectable stage IIIc, IIId and IV melanoma by the American Joint Committee on Cancer (AJCC) (the 8th Edition). (Note: uveal melanoma cases are excluded)
5. Baseline tumor specimens available for NGS analysis or equivalent test results acceptable by the principal investigator.
6. Measurable disease by RECIST v1.1 criteria
7. Adequate organ and marrow function (within 4 weeks prior to study treatment initiation):
8. A negative urine or plasma β-HCG test result is required at screening for female patients of childbearing potential.
9. Contraception is required for patients and their partners throughout the trial and within 1 year after the last dose of study treatment.
10. Capable of understanding and complying with the study protocol requirements ( including follow-up visit and examinations).
11. Be willing to signed a written informed consent document before enrollment.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to recombinant human interferon-α1bcombined, toripalimab and anlotinib hydrochloride.
2. Patients accepted other anti-tumor clinical trials within 4 weeks prior to study entry.
3. Patients accepted anti-tumor radiotherapy within 4 weeks prior to study entry.
4. Disease improved by in response to anti-tumor therapies within 4 weeks including perioperative chemotherapy, molecularly targeted therapy, PD-1/PD-L1/CTLA-4 immune therapy, anti-angiogenesis therapy (such as sunitinib, sorafenib, regorafenib, bevacizumab, imatinib, apatinib) or interferon, herbal supplements.
5. Plan to take other systemic or local anti-tumor therapy during the current study
6. Systemic treatment with either corticosteroid (> 10 mg /kg prednisone equivalents) or other immunosuppressive medications prior to 2 weeks prior to study dose initiation
7. Known hematologic malignancy, primary brain tumor, sarcoma or any other primary solid tumor unless the disease-free period is over 5 years.
8. Imaging confirmed of central nervous system (CNS) metastases with or without meningeal carcinomatosis
9. Known severe hypersensitivity reaction of another mono-antibody therapy.
10. Known active autoimmune disease requiring systemic treatment (such as corticosteroids or immunosuppressive medications) or related replacement therapies (such as thyroid hormone for hypothyroidism, insulin for diabetes or physiological glucocorticoid replacement therapy for adrenal or pituitary insufficiency) in the past 2 years.
11. Individuals with bleeding tendency or under thrombolytic or anticoagulant therapy. Coagulation abnormalities as the following circumstances: INR >1.5；PT > 1.2 ULN；PTT > 1.2 ULN.
12. Use of anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs
13. Obvious hemoptysis or daily hemoptysis above 2.5ml in the past 2 months
14. Any condition has potential risk of gastrointestinal bleeding or perforation, such as active gastrointestinal ulcer, known intra luminal metastases,inflammatory bowel disease; known abdominal fistula, gastrointestinal perforation or intraperitoneal abscess 4 weeks prior to entry of the study entry
15. Open wounds, ulcers or fractures
16. Surgery history within past 4 weeks, except for melanoma removal or partial removal
17. Hereditary or acquired bleeding and thrombotic tendency such as hemophilia, thrombocytopenia, hypersplenism
18. Uncontrolled hypertension defined as persistent systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg despite antihypertension medicine therapy
19. Known cardiovascular diseases as follows in the past 6 months (cerebral vascular accident, transient ischemic attack, cardiac arrhythmia（including QTc ≥ 450 ms for males and QTc ≥ 470 ms for females; angina,coronary angioplasty or coronary stent implantation, pulmonary embolism,untreated deep vein thrombosis or anticoagulation treatment less than six weeks,arterial thrombosis; heart failure patients in NYHA class III and IV; above Ⅱ degrees heart block; myocardial infarction unstable arrhythmia, or unstable angina in the past 6 months; cerebral infarction within 3 months; left ventricular ejection fraction (LVEF) is less than 50% and clinically significant pericardial disease indicated by color doppler echocardiography; ECG indicates acute ischemia or active conduction system abnormalities
20. Use of medications which might lead to Prolonged QT interval and torsades de pointes
21. Other diseases that may affect compliance or interfere with results interpretation including active opportunistic infections or progressing or severe infections , uncontrolled diabetes or pulmonary diseases including interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm. Known HIV or AIDS-related illness, or active HBV, HCV and tuberculosis
22. A history of getting a live vaccine within 4 weeks prior to the first dose; a history of hematopoietic stimulating factor therapy such as colony-stimulating factor (CSF) and erythropoietin (EPO) within 2 weeks prior to the first dose; a history of major surgeon except for diagnosis within 4 weeks prior to the first dose
23. Diagnosis of a psychiatric or substance abuse disorder
24. Individuals who are pregnant or breast-feeding or plan to conceive during the study period
25. Any other illness, laboratory abnormality, or situations that in the opinion of the principal investigator would compromise the patients' ability to tolerate treatment or would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Recommended phase II dose (RP2D) of anlotinib hydrochloride | 12 weeks after first drug administration
  RP2D of anlotinib hydrochloride will be depended according to the dose-limiting toxicities of anlotinib hydrochloride
Phase II: Objective response rate (ORR) | Up to 24 months after the last episode
  proportion of patients with a complete response or partial response to treatment
Phase II: progression-free survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  time from enrollment to progression or death

SECONDARY OUTCOMES:
disease control rate (DCR) | Up to 60 months after the last episode
  the percentage of patients who have achieved complete response, partial response and stable disease to the therapeutic intervention
duration of response (DOR) | Up to 60 months after the last episode
  time from response to progression/death (the earlier event)
overall survival(OS) | From date of enrollment until the date of death from any cause, assessed up to 60 months
  The median and 3 year OS rate of patients with unresectable advanced melanoma treated with the combination regimen of interferon-α1b, toripalimab, and anlotinib hydrochloride
Clinical Benefit Rate(CBR) | Week 0-24
  the proportion of patients with a complete or partial response or with stable disease at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Guannan Zhu, M.D.;Ph.D, Principal Investigator — Xijing Hospital
Locations (1):
- Air Force Military Medical University/ Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided